CLINICAL TRIAL: NCT05053997
Title: NAVIGATE - Improving Survival and Quality of Life in Vulnerable Lung Cancer Patients Through Nurse Navigation, Symptom Monitoring and Exercise: Study Protocol for a Multicenter Randomized Controlled Trial
Brief Title: Navigate - Improving Survival and Quality of Life in Vulnerable Lung Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Danish Cancer Society (Other); Odense University Hospital (Other); Vejle Hospital (Other); Hospital of Southern Jutland (Other)
Responsible Party: Principal Investigator, Susanne Dalton, Professor, MD, PhD, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAVIGATE
Record Dates: First submitted 2021-09-13; First posted 2021-09-23 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAVIGATE intervention arm (Experimental): Nurse navigation
  Interventions: Behavioral: NAVIGATE
- Navigate control arm (No Intervention): Standard treatment and care

INTERVENTIONS:
Behavioral: NAVIGATE — Patients' symptoms are systematically monitored by use of bi-weekly patient reported outcomes and nurse navigators will initiate appropriate actions in terms of medical treatment or guidance of self-management strategies. Nurse navigators will motivate and support patients in health behavior changes and in selfmanaging their treatment and symptoms, and, if relevant, refer to existing rehabilitation services at the hospital or at the local rehabilitation center. Physiotherapists will supervise a training program aimed at improving patients' physical function and thus potentially surgery and overall treatment adherence and outcomes.
  Arms: NAVIGATE intervention arm

SUMMARY:
Half of patients with lung cancer face a limited life span of one-year survival, which is characterized by severe physical and psychological symptoms. Differences in stage, comorbidity but also treatment may explain a large proportion of the social inequality in lung cancer survival. Some vulnerable patients may not receive first line treatment as planned either due to poor performance status or if they are not able to adhere to treatment appointments. Knowing how to navigate the health system may be a barrier preventing vulnerable patients in receiving optimal treatment. The primary aim of this randomised, controlled trial is to test whether a nurse-led individually tailored program including systematic screening of symptoms using PROs and a physical training program will significantly improve a composite outcome of survival and quality of life as the primary outcome among vulnerable lung cancer patients compared with standard care. Secondary outcomes include adherence to cancer treatment, symptom burden and overall survival.

DETAILED DESCRIPTION:
During a period of 3 years and 10 months, consecutive newly diagnosed (< 1 week) lung cancer patients will be pre-screened for eligibility and invited to participate at departments of oncology or respiratory medicine in Denmark. Participants (N=250) will be randomized (1:1) to standard treatment plus the intervention (intervention group) or standard treatment (control group) and followed for 1 year. Patients randomized to the control group will receive standard treatment and care consisting of a nurse and a physician, who sees the patient at treatment schedules and during follow-up, i.e. every 3 months for the first 2 years and subsequently annually up to 5 years.

Data will be collected from the intervention and the control group at baseline within 6 weeks after diagnosis, and 3, 6 months and 12 months after diagnosis. Physical tests will be performed at baseline and after 3 and 6 months. Baseline physical tests will be allowed after randomization if patients have difficulties in attending the physiotherapy department within 6 weeks after their diagnosis. Considering that participating patients are vulnerable with limited resources we will proactively support patients in responding to questionnaires electronically, on paper or via telephone as per patient's preference allowing evaluation of the primary and secondary outcomes as well as covariates and mechanisms. The treatment factors will be obtained from the lung cancer clinical database and individual medical journals. In order to develop cost utility analyses, information on use of health services will be retrieved from the national registers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Diagnosed with NSCLC at all stages regardless of treatment intension at the participating departments
* Performance status ≤ 2
* Vulnerable according to pre-defined criteria

Exclusion Criteria:

* Severe untreated psychiatric disorder (e.g. psychosis) or cognitive problems (e.g. dementia) preventing informed consent
* Not able to receive treatment
* Not able to read and understand Danish -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
A hierarchical composite outcome of survival and global quality of life | 3 months from randomization
  Measured from death from all causes and the Global Health Status (a subscale of EORTC QLQ-C30)

SECONDARY OUTCOMES:
Overall survival | 3 months from randomization
  Measured by death from all causes
Overall survival | 6 months from randomization
  Measured by death from all causes
Overall survival | 12 months from randomization
  Measured from death from all causes
Adherence to cancer treatment | 3 months from randomization
  Measured by date of skipped treatments or delays if any, and dose administered
Adherence to cancer treatment | 6 months from randomization
  Measured by date of skipped treatments or delays if any, and dose administered
Adherence to cancer treatment | 12 months from randomization
  Measured by date of skipped treatments or delays if any, and dose administered
Symptom burden and health related quality of life | 3 months from randomization
  Measured by EORTC Questionnaire Core 30 (QLQ-C30) and the lung module (QLQ-LC13).
  The QLQ-C30 questionnaire consists of 30 questions with five functional scales (physical, role, cognitive, emotional and social), three symptom scales, a global health status / QoL scale, and six single items.
  The QLQ-LC13 module comprises both multi-item and single-item measures of lung cancer-associated symptoms (coughing, haemoptysis, dyspnoea and pain) and side-effects from conventional chemo- and radiotherapy (hair loss,neuropathy, sore mouth and dysphagia).
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Symptom burden and health related quality of life | 6 months from randomization
  Measured by EORTC Questionnaire Core 30 (QLQ-C30) and the lung module (QLQ-LC13).
  The QLQ-C30 questionnaire consists of 30 questions with five functional scales (physical, role, cognitive, emotional and social), three symptom scales, a global health status / QoL scale, and six single items.
  The QLQ-LC13 module comprises both multi-item and single-item measures of lung cancer-associated symptoms (coughing, haemoptysis, dyspnoea and pain) and side-effects from conventional chemo- and radiotherapy (hair loss, neuropathy, sore mouth and dysphagia).
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Symptom burden and health related quality of life | 12 months from randomization
  Measured by EORTC Questionnaire Core 30 (QLQ-C30) and the lung module (QLQ-LC13).
  The QLQ-C30 questionnaire consists of 30 questions with five functional scales (physical, role, cognitive, emotional and social), three symptom scales, a global health status / QoL scale, and six single items.
  The QLQ-LC13 module comprises both multi-item and single-item measures of lung cancer-associated symptoms (coughing, haemoptysis, dyspnoea and pain) and side-effects from conventional chemo- and radiotherapy (hair loss,neuropathy, sore mouth and dysphagia).
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Quality of life (QOL) measured by EuroQol EQ-5D-5L | 3 months from randomization
  EQ-5D-5L measures individual generic health status using 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and each dimension has 5 levels depending on severity of symptoms (1 no problems, 5 extreme problems) and a VAS (visual analogue scale). The scores can then be converted into a single index number. The index value will be used for calculation of quality-adjusted life years (QALYs) for a health economic analysis of the intervention.
Quality of life (QOL) measured by EuroQol EQ-5D-5L | 6 months from randomization
  EQ-5D-5L measures individual generic health status using 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and each dimension has 5 levels depending on severity of symptoms (1 no problems, 5 extreme problems) and a VAS (visual analogue scale). The scores can then be converted into a single index number. The index value will be used for calculation of quality-adjusted life years (QALYs) for a health economic analysis of the intervention.
Quality of life (QOL) measured by EuroQol EQ-5D-5L | 12 months from randomization
  EQ-5D-5L measures individual generic health status using 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and each dimension has 5 levels depending on severity of symptoms (1 no problems, 5 extreme problems) and a VAS (visual analogue scale). The scores can then be converted into a single index number. The index value will be used for calculation of quality-adjusted life years (QALYs) for a health economic analysis of the intervention.
Health behavior | 3 months from randomization
  Measured by single-items questions related to physical activity, alcohol consumption and smoking behavior
Health behavior | 6 months from randomization
  Measured by single-items questions related to physical activity, alcohol consumption and smoking behavior.
Health behavior | 12 months from randomization
  Measured by single-items questions related to physical activity, alcohol consumption and smoking behavior.
Self-efficacy and self-activation | 3 months from randomization
  Measured by single items from Patient Activation Measure (PAM) and Health Education Impact Questionnaire (HEIQ)
Self-efficacy and self-activation | 6 months from randomization
  Measured by single items from Patient Activation Measure (PAM) and Health Education Impact Questionnaire (HEIQ)
Self-efficacy and self-activation | 12 months from randomization
  Measured by single items from Patient Activation Measure (PAM) and Health Education Impact Questionnaire (HEIQ)
Rehabilitation services | 3 months from randomization
  Measured by single item question
Rehabilitation services | 6 months from randomization
  Measured by single item question
Rehabilitation services | 12 months from randomization
  Measured by single item question
Process evaluation | 3 months from evaluation
  Evaluation by participant-observations during training and patient sessions with subsequent qualitative semi-structured interviews with participants about their experience of the intervention components; however, only among participants who provide informed consent for this. Focus group interviews with nurse navigators and physiotherapists will be conducted about their perceptions of the intervention (facilitators and barriers).
  Additionally, evaluation of intervention components will be measured using quantitative single-items questions
Process evaluation | 12 months from evaluation
  Evaluation by participant-observations during training and patient sessions with subsequent qualitative semi-structured interviews with participants about their experience of the intervention components; however, only among participants who provide informed consent for this. Focus group interviews with nurse navigators and physiotherapists will be conducted about their perceptions of the intervention (facilitators and barriers).
  Additionally, evaluation of intervention components will be measured using quantitative single-items questions.
Cost-effectiveness | 12 months from randomization
  Evaluation by health care costs and QALYs (Quality Adjusted Life Years) between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne O Dalton, Professor, Principal Investigator — Zealand University Hospital; Pernille E Bidstrup, PhD, Principal Investigator — Danish Cancer Society; Erik Jakobsen, PhD, Principal Investigator — The Danish Lung Cancer Research Center
Locations (6):
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Gødstrup Hospital, Herning
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde
  - Sønderborg Sygehus, Sønderborg
  - Vejle Sygehus, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Langballe R, Svendsen L, Jakobsen E, Dalton SO, Karlsen RV, Iachina M, Freund KM, Leclair A, Jorgensen LB, Skou ST, Ehlers JH, Torenholt R, Svendsen MN, Envold Bidstrup P. Nurse navigation, symptom monitoring and exercise in vulnerable patients with lung cancer: feasibility of the NAVIGATE intervention. Sci Rep. 2023 Dec 20;13(1):22744. doi: 10.1038/s41598-023-50161-w. PMID 38123657
- [Derived] Langballe R, Dalton SO, Jakobsen E, Karlsen RV, Iachina M, Freund KM, Leclair A, Nielsen AS, Andersen EAW, Rosthoj S, Jorgensen LB, Skou ST, Bidstrup PE. NAVIGATE: improving survival in vulnerable patients with lung cancer through nurse navigation, symptom monitoring and exercise - study protocol for a multicentre randomised controlled trial. BMJ Open. 2022 Oct 31;12(10):e060242. doi: 10.1136/bmjopen-2021-060242. PMID 36316074

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-12-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT05053997/SAP_000.pdf